CLINICAL TRIAL: NCT06813820
Title: RELIVE (Randomized Evaluation of Less Invasive Ventricular Enhancement) Trial
Acronym: RELIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioVentrix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0100
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Left Ventricle Remodeling; Left Ventricle Dilated; CHF
Keywords: Left Ventricle Reverse remodeling
MeSH Terms: conditions — Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Revivent System Therapy plus Guideline Directed Medical Therapy (GDMT) (Experimental): Medical Intervention through a mini thoracotomy, placement of anchors to plicate the scarred areas of the heart thereby reducing the left ventricle size and improving left ventricle mechanics. Subjects would continue on Guideline Directed Medical Therapy (GDMT)
  Interventions: Device: Revivent System
- Guideline Directed Medical Therapy (GDMT) only (No Intervention): Subjects would remain on Guideline Directed Medical Therapy (GDMT) with no additional medical intervention.

INTERVENTIONS:
Device: Revivent System — BioVentrix has developed the Revivent System to mirror Surgical Ventricular Restoration (SVR). The Revivent System is used to place permanent cardiac implants to the epicardial surface for the purpose of reconfiguring abnormal cardiac geometry that is contributing to the dysfunction.
  Arms: Revivent System Therapy plus Guideline Directed Medical Therapy (GDMT)

SUMMARY:
A prospective, multi-center randomized trial comparing the Revivent System plus GDMT to GDMT alone. A total of approximately 135 subjects will be randomized in a 2:1 allocation ratio (90 treatment and 45 control), with approximately 128 evaluable patients and assuming 5% loss to follow-up. A primary safety endpoint will be evaluated at 30 days. Primary efficacy endpoint will be at 1 year. Interim efficacy endpoints will be evaluated at 6 months.

DETAILED DESCRIPTION:
The purpose of the study is to assess the safety and effectiveness of the BioVentrix Revivent System plus GDMT compared to GDMT alone for the treatment of LV anterior/apical scar/aneurysm with possible additional involvement of the lateral, septal, and/or inferior regions in patients with symptomatic heart failure.

Safety will be assessed compared with a Performance Goal based on surgical ventriculoplasty outcomes (MAE's at 30 days).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. LV Aneurysm or Scar Presence: Defined by presence of a contiguous acontractile (akinetic and/or dyskinetic) non-calcified scar
3. LV Aneurysm/Scar Location: Defined as a scar involving anterior, apical or anterolateral ± septal regions of the left ventricle as evidenced by cardiac imaging (Viability of myocardium in regions remote from area of intended scar exclusion as evidenced by cardiac imaging)
4. Left Ventricular Ejection Fraction < 40%
5. Left ventricular end-systolic volume index ≥60 mL/m2
6. Suffering from heart failure symptoms as defined by NYHA Classification > 2 not responsive to medical therapy
7. Patient completed 6 Minute Walk Test and KCCQ Quality of Life Questionnaire (can be performed at baseline visit)
8. Patient is on adequate Guideline Directed Medical Therapy (GDMT)
9. Subject or a legally authorized representative must provide written informed consent
10. Agree to required follow-up visits
11. Female subject of childbearing potential does not plan pregnancy for at least one year following the index procedure. For a female of childbearing potential, a pregnancy test must be performed with negative results known within seven days prior to index procedure

Exclusion Criteria:

Candidates will be excluded from the study if ANY of the following conditions is present:

1. Cardiac Resynchronization Therapy (CRT) or ICD pacing lead placement ≤ 90 days prior to enrollment
2. Valvular heart disease, which in the opinion of the investigator, will require intervention (transcatheter or surgical)
3. Mitral Regurgitation greater than moderate (>2+)
4. Need for coronary revascularization, in the opinion of the investigator
5. Peak Systolic Pulmonary Arterial Pressure > 70 mm Hg via echo or right heart catheterization
6. Myocardial Infarction within 90 days prior to enrollment
7. Within the last six months, a prior CVA or TIA, or intracranial hemorrhage
8. Co-morbid disease process with life expectancy of less than one year or active malignancy not in remission
9. Severe pulmonary disease that would preclude general anesthesia
10. Any solid organ transplant or is on waiting list for any solid organ transplant other than cardiac
11. Chronic renal failure with a GFR<30ml/min
12. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events Composite Performance Goal | 30 days
  Composite of Major Adverse Events at 30 days comprised of Clinical Events Committee (CEC) Adjudication of Mortality, Myocardial Infarction (MI), Major Stroke, Prolonged Intubation >48hrs, Need for Inotropic support >24hrs, Mech circulatory support intra or post op, BARC 4 or 5 bleeding, reoperation, serious infection related to device or procedure, Cardiac tamponade, or Initiation of renal replacement therapy, with a Performance Goal (PG) of 70% (upper bound of the 97.5% one sided CI)
Composite Effectiveness Endpoint | 6 Months
  Using Finkelstein Schoenfeld (FS) hierarchical approach. This approach compares each treatment subject versus each control subject in a hierarchal fashion beginning with Kansas City Cardiomyopathy Questionnaire (+10 point improvement with higher score being better), 6 Minute Walk Test (+25meter improvement with longer distance being better), change in New York Heart Association (NYHA) Class (+1 point improvement with scale being 1 to 4 with lower value being better). Begin comparing at highest hierarchal assessment. If one group is "better than" the other, count as "win". If treatment and control subject equal at that assessment, compare to next hierarchal measure, if equal again, go to next until you have a "win". Compare overall wins versus loses for an overall win ratio.
Composite Effectiveness Endpoint | 12 Months
  Using Finkelstein Schoenfeld (FS) hierarchical approach - Cardiovascular Mortality, Heart Transplant, Left Ventricular Assist Device (LVAD) Implantation, Hospital Readmission, Kansas City Cardiomyopathy Questionnaire (+10 point improvement with higher score being better), 6 Minute Walk Test (+25meter improvement with longer distance being better), change in New York Heart Association (NYHA) Class (+1 point improvement with scale being 1 to 4 with lower value being better). Begin comparing at highest hierarchal assessment. If one group is "better than" the other, count as "win". If treatment and control subject equal at that assessment, compare to next hierarchal measure, if equal again, go to next until you have a "win". Compare overall wins versus loses for an overall win ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod THourani, MD, Principal Investigator — Piedmont Healthcare; Marat Fudim, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Penn State Health, Hershey, Pennsylvania